CLINICAL TRIAL: NCT04479228
Title: A Randomized Control Trial of Plastic Stents vs. NAGI Bi-flanged Metal Stent for Endoscopic Ultrasound Guided Drainage of Walled-off Necrosis
Brief Title: Plastic Stents vs. NAGI Bi-flanged Metal Stent for Endoscopic Ultrasound Guided Drainage of Walled-off Necrosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WON_NAGIvsPlastic
Record Dates: First submitted 2020-07-15; First posted 2020-07-21 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Acute Necrotizing Pancreatitis; Walled Off Necrosis
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NAGI bi-flanged metal stent (BFMS) (Experimental): The WON will be punctured using a standard 19-gauge FNA needle and the aspirate was sent for biochemical and microbial analysis. A 0.025-inch (Visiglide; Olympus Corporation, Tokyo, Japan) or 0.035-inch stiff guidewire (Jag Wire; Boston Scientific) passed through the needle into the cyst cavity to form at least 1 to 2 loops under fluoroscopic guidance. A 6F cystotome (Endo-flex GmbH Dusseldorf, Germany) will be passed over the guidewire for creating a fistula. Subsequently, a 6-mm balloon dilator (Hurricane; Boston Scientific Corporation or Titan balloon, Wilson Cook) will be used to further dilate the fistula tract. After this, the stent delivery catheter is advanced over the guidewire across the PFC wall and the BFMS (Nagi; Taewoong Medical, Gyeonggi-do, South Korea) deployed using sonographic, fluoroscopic and endoscopic visualization.
  Interventions: Device: Endosonography guided transmural drainage
- Plastic stents (Experimental): Double-pigtail plastic stents will be used. A minimum of one 10Fr pigtail plastic stent will be placed. After initial EUS-guided access, the ostomy will be dilated first, using a cystotome, and secondly with a balloon dilation. The plastic stent will be inserted and delivered following the routine technique of each interventional endoscopist. The number of the plastic stents and the size of the balloon used to dilate the ostomy will depend on the WON size and content.
  Interventions: Device: Endosonography guided transmural drainage

INTERVENTIONS:
Device: Endosonography guided transmural drainage — The procedures would be performed by experienced endoscopists. All procedures will be performed with the patient in the left lateral position under propofol sedation after administration of intravenous antibiotics (third generation cephalosporins) A therapeutic linear echo-endoscope (UCT-180; Olympus Ltd, Tokyo, Japan) will be used; the PFC assessed for size, wall maturity, thickness, interposing collaterals and percentage of solid debris

SUMMARY:
Introduction:

Walled off necrosis (WON) is defined as a well circumscribed pancreatic and/or peri pancreatic necrosis containing a variable amount of necrotic tissue. WON usually occurs >4 weeks after onset of necrotizing pancreatitis. It is associated with significant morbidity and mortality especially if infected. Symptomatic WON should be drained either percutaneously, endoscopically or surgically. Minimal invasive approaches are being increasingly used for effective management of WON as it is associated with less adverse events. Various recent studies have shown that endoscopic approach have improved clinical outcome, less hospital stay and lower cost compared to surgical approach.

Endoscopic ultrasound guided drainage of WON with either plastic stents or lumen apposing metal stents (LAMS) is mainstay of WON management. A systemic review based on retrospective comparative studies showed no difference regarding treatment success for WON by plastic or metal stents6. However, metal stent had shorter procedure time. A Single center RCT from USA comparing LAMS vs multiple plastic stents for WON has shown that except shorter procedure duration, there was no significant difference in treatment outcomes. To minimize LAMS related adverse events, it should be removed within 3 weeks. However, in the same study 25.8% patients of LAMS group and 55.2% patients of plastic stent group underwent additional intervention within 72 hours for persistent symptoms.

Larger diameter, specific stent designs to reduce adverse events should have better outcome with LAMS as compared to plastic stents. Primary outcome of this single center randomized controlled trial is to examine whether dedicated NAGI bi-flanged metal stents (BFMS) are superior to plastic stent in terms of short term and long term success.

Aims and Hypothesis:

The aim of the current study is to study whether NAGI BFMS are superior to plastic stent in terms of short term and long term success in the EUS guided drainage of WON.

The investigators hypothesize that the clinical success with NAGI BFMS would be better than plastic stents in the EUS guided drainage of WON.

DETAILED DESCRIPTION:
1.1 Patient recruitment Patients would be recruited from the in-patient or outpatient department prior to their scheduled endoscopic intervention.

1.2 Study design This is a single center randomized controlled study with two parallel groups without masking with a 1:1 allocation ratio

1.3. Study intervention - stent placement The procedures would be performed by experienced endoscopists. All procedures will be performed with the patient in the left lateral position under propofol sedation after administration of intravenous antibiotics (third generation cephalosporins) A therapeutic linear echo-endoscope (UCT-180; Olympus Ltd, Tokyo, Japan) will be used; the PFC assessed for size, wall maturity, thickness, interposing collaterals and percentage of solid debris.

NAGI BFMS - The WON will be punctured using a standard 19-gauge FNA needle and the aspirate was sent for biochemical and microbial analysis. A 0.025-inch (Visiglide; Olympus Corporation, Tokyo, Japan) or 0.035-inch stiff guidewire (Jag Wire; Boston Scientific) passed through the needle into the cyst cavity to form at least 1 to 2 loops under fluoroscopic guidance. A 6F cystotome (Endo-flex GmbH Dusseldorf, Germany) will be passed over the guidewire for creating a fistula. Subsequently, a 6-mm balloon dilator (Hurricane; Boston Scientific Corporation or Titan balloon, Wilson Cook) will be used to further dilate the fistula tract. After this, the stent delivery catheter is advanced over the guidewire across the PFC wall and the BFMS (Nagi; Taewoong Medical, Gyeonggi-do, South Korea) deployed using sonographic, fluoroscopic and endoscopic visualization.

Plastic stents - Double-pigtail plastic stents will be used. A minimum of one 10Fr pigtail plastic stent will be placed. After initial EUS-guided access, the ostomy will be dilated first, using a cystotome, and secondly with a balloon dilation. The plastic stent will be inserted and delivered following the routine technique of each interventional endoscopist. The number of the plastic stents and the size of the balloon used to dilate the ostomy will depend on the WON size and content.

1.4 Stents NAGI bi-flanged metal stent (BFMS)- Nagi stent is a dedicated self-expandable fully covered bi-flanged metal stent (BFMS) for drainage of pancreatic fluid collections. The stent is short in length (20 or 30 mm) with caliber (10, 12, 14, or16 mm) having flared ends (diameter 26 mm). Procedure-related adverse events will be managed accordingly and documented Plastic stents - Two 7fr or 10 fr plastic stents will be used 1.5 Randomization The patients would be randomised will be randomised to Plastic vs NAGI BFMS by using Med Cal C software (version 12.3, Belgium). There will be no masking.

1.6 Post-procedural management After the drainage procedure, patients will be observed in the hospital for symptomatic improvement or development of any adverse events. Oral liquids are allowed 6 hours after the procedure. Intravenous antibiotics will be continued for 2 to 3 days which will be later changed to the oral route.

All patients will be re-assessed within 72 hours after EUS guided drainage for symptomatic relief. In case of persistent symptoms, the most beneficial therapeutic approach for the patient will be adopted as per expert multimodality team of endoscopists, surgeon and interventional radiologist such as placement of nasocystic drain, coaxial plastic stent placement in BFMS, endoscopic necrosectomy or percutaneous drainage.

In case of symptomatic relief and significant reduction in size of WON, patient will be followed up after 1 week and at 4 week or early if symptoms recur and/or any new symptom appears. In case of complete symptomatic relief and disappearance of WON at 4 weeks, metal stent will be removed.

If persistent collection or there is evidence of DPDS, then in patients with initial plastic stent placement, stent will not be removed. In BFMS group, BFMS will be replaced by plastic stent. Patient will be observed in hospital for 24 hours 1.7 Outcome measurements The primary outcome measurement is Clinical success at 4 weeks determined by the reduction of the collection (<50% or <5 cm in size) along with resolution of symptoms Secondary outcomes include

1. Re-interventions
2. Long term clinical success at 24 weeks
3. Adverse events
4. Cost - effectiveness

Technical success: It is defined as the correct deployment of stent at both ends with visualization of drainage of the liquid.

Clinical success: It is defined as resolution of symptoms and significant reduction in of collection size (< 50% or <5 cm in size).

Recurrence: It is appearance of symptomatic fluid collection evident on imaging during follow-up after documented clinical success.

Adverse events: It is defined as undesirable situations during the study period whether related or unrelated to the EUS guided drainage.

1.8 Follow-up Patient will be assessed on day 1 to 3, then at 1, 4, 8 weeks followed by 12 and 24 weeks by personnel participating in the study. At each visit, information regarding signs and symptoms, adverse events and recurrence will be collected. In case of mortality during study period, any possible relation to endoscopic procedure will be investigated and will be noted.

1.9 Sample size calculation The success rate of metal stent is assumed as 75 % and 45% for plastic stent. The required sample size with 80% power and 0.05 as type 1 error is 40 per group

Statistical Formula for estimation of sample size :

n= 2 (Zα +Zβ)2 (P1+Q1+P2+Q2)/ (P1 -P2 ) X(P1-P2)

where, n = Sample size

P1 proportion of outcome measure under Group1 (Success rate of metal stent and assumed to be 75 %) Q1 proportion of failure rate metal stent (1 - 0.85 ) P2 proportion of success rate in plastic group2 (success rate and assumed as 45 %) Q2 proportion failure rate of plastic stent in group 2 (1 - 0.45) zα is factor corresponding to type 1 error with two sided test and is taken as 1.96 Zβ factor corresponding to type 11 error i.e (1- β) is power of and is usually taken as 80 % and the value =0.84 Forty patients will be recruited in each group to reject the null hypothesis that the proportion of clinical success in the LAMS group is equal to that of the plastic stent group with an 80% power with 5% type 1 error. A planned interim analysis will be done at half of the recruitment.

1.10 Statistical analyses The continuous variables will be described as mean, standard deviation, median, range and interquartile range. Categorical variables will be described as percentages of different categories.

Primary outcome will be tested with chi-square test or Fisher's exact test. The level of significance has been set at 5%. To quantify the magnitude of the difference the relative risk and odds ratio will be calculated with 95% confidence interval. Univariate and multivariate analysis will be done to determine which are the factors associated with clinical success and clinical recurrence. Kaplan-Meier survival analysis will be done for appearance clinical recurrence.

1.11 Withdrawal of individual subjects Subjects can leave the study at any time for any reason if they wish to do so without any consequences. The treating physician can decide to withdraw a subject from the study for any medical reason. In case of withdrawal, the reason for withdrawal and, if applicable, the alternative treatment, would be recorded.

1.12 Participating centres Asian Institute of Gastroenterology - Hyderabad

ELIGIBILITY:
Inclusion Criteria:

* Adult >18 years,
* Patient with symptomatic WON
* Debris <50% (based on cross sectional imaging)
* Written informed consent

Exclusion Criteria:

* Pregnancy or breast feeding,
* Severe coagulopathy INR >1.5 which is not correctable and/or platelets <50000/mm3
* Endoscopic drainage is technically not feasible
* Fluid collections other than WON
* Patient who is unable to understand study protocol or not willing for follow-up requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2021-08-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of patient achieving Clinical Success | 4 weeks
  Clinical success at 4 weeks determined by the reduction of the collection (<50% or <5 cm in size) along with resolution of symptoms.

SECONDARY OUTCOMES:
Re-Interventions | 4 weeks
  The number of re-interventions required to achieve primary outcome, which includes need for necrosectomy, nano-cystic drainage placement, placement for nasogastric or nasojejunal tube for feeding, need for percutaneous or surgical drainage.
Number of patients achieving Long term success | 24 weeks
  Long term success defined as absence of persistent collection or recurrence at 24 weeks.
Number of patients developing Adverse events | 24 weeks
  It is defined as undesirable situations during the study period whether related or unrelated to the EUS guided drainage.

IPD SHARING:
Plan to Share IPD: No
Data sharing won't be allowed to outside researcher.